CLINICAL TRIAL: NCT03717090
Title: Rapid Diagnosis of Prosthetic Joint Infection by Matrix-assisted Laser Desorption Ionization Time-of-flight Mass Spectrometry
Brief Title: Rapid Diagnosis of Prosthetic Joint Infection by Matrix-assisted Laser Desorption
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Feng Chih Kuo, Assistant professor, Chang Gung Memorial Hospital
Other Study IDs: CMRPG8F1402
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Prosthetic Joint Infection
Keywords: mass spectrometry, diagnosis, prosthetic joint infection, matrix-assisted laser desorption ionization
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PJI
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Sample collection study Sample collection and collection of laboratory values

SUMMARY:
This is a prospective cohort study. All patients presenting for periprosthetic joint infection and requiring debridement only or resection arthroplasty will be eligible. The synovial joint fluid will be sampled before the arthrotomy at the operation room.

The purpose of this study will be to evaluate that 1) the concordance of organism identification by the direct identification of MALTI-TOF MS versus routine identification of MALTI-TOF MS and conventional cultures and 2) the timing of preliminary strain identification by the direct identification of MALTI-TOF MS, routine identification of MALTI-TOF MS and conventional cultures in patients with periprosthetic joint infection.

DETAILED DESCRIPTION:
Material and Methods

1. Patients who have a high probability of infection based on the Musculoskeletal Infection Society (MSIS) criteria and are scheduled for debridement only or debridement with implant removal, will be invited to enroll the study after signed informed consent.

   The synovial joint fluid will be sampled before the arthrotomy at the operation room. Aspirates will be collected under an aseptic technique with an 18-Fr sterile syringe with a minimum amount of 14 ccs. The sample will be divided between MALDI-TOF mass spectrometry in standard blood culture bottles (10 ccs), wound culture tube (2 ccs), and synovial fluid analysis (2 ccs). The samples will be delivered to microbiology laboratory within a 2-hour period.
2. Bacterial culture and conventional identification Bacterial identification will be performed by the conventional method using the Vitek 2 system. For the conventional culture, 1 µL of well-mixed synovial joint fluid will be inoculated and spread onto blood agar plates and MacConkey agar plates using a sterile plastic disposable loop. Plates will be incubated in an aerobic atmosphere at 37℃ for 18-24 hr. When bacterial growth is observed, the colonies on blood agar will be counted, and colonies from both types of plates will be identified by using the Vitek 2 system.
3. MALDI-TOF MS identification The suspension obtained following the above sample preparation will be centrifuged at 13,000g for 2 minutes, and the supernatant will be discarded. The pellet will be centrifuged at 13,000g for another 2 minutes prior to the removal of the residual ethanol. Fifty microliters of formic acid (70% v/v) and 50 mL of 100% acetonitrile will be added to the pellet, and mixed thoroughly after each reagent is added. The suspension will be centrifuged again at 13,000g for another 2 minutes, and 1 mL of the supernatant will be spotted onto the steel target plate. Analysis will be performed following air-drying of 1 mL a-cyano-4-hydroxycinnamic acid matrix solution placed onto the dried sample spot in duplicate.

   Mass spectra profiles will be acquired using a microflex LT MALDI-TOF mass spectrometer (Bruker Daltonics, Bremen, Germany) following the manufacturer's settings. Spectra will be recorded in the linear positive mode at a laser frequency of 60 Hz within a mass range from 2000 Da to 20,000 Da. All bacteria identifications will be performed by MALDI-TOF Biotyper RTC and the Bruker MALDI Biotyper 3.1 software and library (4613 isolates; Bruker Daltonics). Criteria used for microorganism analysis and identification will be as recommended by the manufacturer.
4. Statistical analysis Time to identification will be determined as the time from colony formation to the time at which the final result is reported to a physician. Statistical analysis will be performed to compare the three methods using Chi-square tests. The level of statistical significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria: high probability of infection based on the Musculoskeletal Infection Society (MSIS) criteria and will be scheduled for debridement only or debridement with implant removal

Exclusion Criteria:

* Patients not meeting MSIS criteria
* Patients undergoing aseptic revision
* Insufficient synovial fluid amount for analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The synovial joint fluid will be sampled before the arthrotomy at the operation room. Aspirates will be collected under an aseptic technique with an 18-Fr sterile syringe with a minimum amount of 14 cc. The sample was partitioned between two set of aerobic and anaerobic BCBs (at least 2.5cc for each bottle), wound culture tube (2cc), synovial fluid analysis (2cc). In instances where there is insufficient fluid to send all 3 modalities (less than 14 mL), patients will be excluded from the current investigation. Samples will be delivered to the clinical microbiology laboratory within a 2-hour period.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
The identification rate of microorganisms | Immediate post-operative period (usually within 5-7 days following surgery)
  The organism identification from direct identification of MALTI-TOF MS, routine identification of MALTI-TOF MS and conventional cultures

SECONDARY OUTCOMES:
The timing of organism identification | Immediate post-operative period (usually within 5-7 days following surgery)
  The timing of preliminary strain identification of direct identification of MALTI-TOF MS, routine identification of MALTI-TOF MS and conventional cultures

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Chih Kuo, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peersman G, Laskin R, Davis J, Peterson M. Infection in total knee replacement: a retrospective review of 6489 total knee replacements. Clin Orthop Relat Res. 2001 Nov;(392):15-23. PMID 11716377
- [Background] Fink B, Makowiak C, Fuerst M, Berger I, Schafer P, Frommelt L. The value of synovial biopsy, joint aspiration and C-reactive protein in the diagnosis of late peri-prosthetic infection of total knee replacements. J Bone Joint Surg Br. 2008 Jul;90(7):874-8. doi: 10.1302/0301-620X.90B7.20417. PMID 18591595
- [Background] Geller JA, MacCallum KP, Murtaugh TS, Patrick DA Jr, Liabaud B, Jonna VK. Prospective Comparison of Blood Culture Bottles and Conventional Swabs for Microbial Identification of Suspected Periprosthetic Joint Infection. J Arthroplasty. 2016 Aug;31(8):1779-83. doi: 10.1016/j.arth.2016.02.014. Epub 2016 Feb 24. PMID 27020677
- [Background] Peel TN, Dylla BL, Hughes JG, Lynch DT, Greenwood-Quaintance KE, Cheng AC, Mandrekar JN, Patel R. Improved Diagnosis of Prosthetic Joint Infection by Culturing Periprosthetic Tissue Specimens in Blood Culture Bottles. mBio. 2016 Jan 5;7(1):e01776-15. doi: 10.1128/mBio.01776-15. PMID 26733067
- [Background] Croxatto A, Prod'hom G, Greub G. Applications of MALDI-TOF mass spectrometry in clinical diagnostic microbiology. FEMS Microbiol Rev. 2012 Mar;36(2):380-407. doi: 10.1111/j.1574-6976.2011.00298.x. Epub 2011 Aug 22. PMID 22092265
- [Background] Haiko J, Savolainen LE, Hilla R, Patari-Sampo A. Identification of urinary tract pathogens after 3-hours urine culture by MALDI-TOF mass spectrometry. J Microbiol Methods. 2016 Oct;129:81-84. doi: 10.1016/j.mimet.2016.08.006. Epub 2016 Aug 5. PMID 27503535